CLINICAL TRIAL: NCT06525259
Title: DISCOVERY of Risk Factors for Type 2 Diabetes in Youth
Acronym: DISCOVERY
Status: Recruiting | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Barbara Braffett, Associate Professor, George Washington University
Other Study IDs: U01DK134971 (NIH)
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus Type 2, Childhood-Onset
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of the DISCOVERY study is to provide innovative critical information regarding the unique natural history of glycemic control, insulin sensitivity, and β-cell function, and their mechanistic determinates, in obese adolescents at risk for developing type 2 diabetes.

DETAILED DESCRIPTION:
The DISCOVERY study will extensively phenotype a large cohort of youth at-risk for type 2 diabetes, as they transition through puberty, and characterize the course of dysfunction in pathophysiological indicators that lead to type 2 diabetes. The knowledge gained from this study of the pathophysiology and epidemiology of youth-onset type 2 diabetes with deep biochemical, clinical, and psychosocial phenotyping will critically inform the design and testing of future treatment and prevention approaches.

ELIGIBILITY:
Inclusion Criteria:

Screening will occur to enrich the yield of individuals who are highly predisposed to develop youth-onset type 2 diabetes and include those with all of the criteria in Category A:

* Overweight or obesity with BMI ≥85th percentile
* Age 9-13 year for girls, 10-14 year for boys (inclusion younger for girls as puberty tends to start a year earlier in girls)
* Tanner Stage 2, 3, or 4
* Elevated HbA1c 5.5-6.4%

Participants who meet all of these categories will further need to meet at least one criterion in Category B:

* Family history of type 2 diabetes in 1st or 2nd degree relative
* Personal exposure to maternal diabetes (i.e., gestational diabetes mellitus (GDM) or mother with type 1 or type 2 diabetes while pregnant with participant)
* HbA1c ≥6.0%
* Severe obesity (BMI ≥99th percentile)
* Personal history of intrauterine growth restriction (IUGR), small for gestational age (SGA), or low birth weight

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation:

* Diabetes based on history, or HbA1c ≥6.5% in the medical record or at screening
* Unable/unwilling to provide consent/participate fully
* Conditions predisposing to diabetes or altering the trajectory of puberty (transplant, cancer, Down Syndrome, Turner Syndrome, Klinefelter Syndrome, ovarian/testicular failure, etc.)
* Medications affecting glucose dynamics during the screening and enrollment period (oral steroids, inhaled steroids >1,000mcg/day past month, atypical antipsychotics, topiramate)
* Prior treatment with insulin
* Use of glucagon-like peptide-1 (GLP-1) receptor agonist or any weight loss medications in the 6 weeks prior to enrollment
* Planning treatment with glucagon-like peptide-1 (GLP-1) receptor agonist or any weight loss medications
* Use of metformin or any glucose lowering medication for a reason other than treatment of diabetes (e.g., for PCOS) in the 6 weeks prior to enrollment
* Known syndromic/monogenic obesity
* Blood disorders impacting HbA1c (e.g., anemia, hemoglobin variants)
* Major systemic organ disease
* History of bariatric surgery or currently planning bariatric surgery
* Current pregnancy or currently planning pregnancy
* Use of GnRH agonist, estrogen, or testosterone
* Individuals who do not speak English or Spanish, given validation of the questionnaires to be utilized

Ages: 9 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: 3,600 youth, aged 9-14 years at enrollment, of all genders and race/ethnic groups from 15 clinical centers in the United States will be included. Youth will be overweight or obese (BMI ≥85th percentile for age) and have evidence of dysglycemia with an HbA1c range from 5.5-6.4% at screening.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Type 2 diabetes | Through study completion, an average of 2.5 years
  Development of type 2 diabetes, as defined by a hemoglobin A1c (HbA1c) ≥6.5% at an annual or mid-year visit followed by a confirmatory HbA1c ≥6.5% collected within 2 weeks of the first value.

SECONDARY OUTCOMES:
Glycemia, β-cell function, insulin sensitivity, and free fatty acid flux | Through study completion, an average of 2.5 years
  Intermediary changes in glycemia, β-cell function, insulin sensitivity, and free fatty acid flux along the spectrum of normal glycemia to prediabetes to type 2 diabetes.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona State University, Phoenix, Arizona
  - Phoenix Children's, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Children's/Joslin Diabetes Center/Massachusetts General Hospital, Boston, Massachusetts
  - Colorado Navajo Nation, Shiprock, New Mexico
  - NYU Langone Health- Brooklyn, Brooklyn, New York
  - NYU Langone Health- Long Island, Garden City, New York
  - NYU Langone Health- Manhattan, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Atrium Health, Charlotte, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine / Texas Children's, Houston, Texas

IPD SHARING:
Plan to Share IPD: No